CLINICAL TRIAL: NCT00652509
Title: Journey for Control of Diabetes Study
Brief Title: Journey for Control of Diabetes Study (0431-111)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 0431-111; 2008_510
Record Dates: First submitted 2008-03-31; First posted 2008-04-03 (Estimated); Last update posted 2017-04-28 (Actual); Status verified 2017-04

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2

ARMS (3):
- 1 (Experimental): IDEA
  Interventions: Behavioral: Interactive Dialogue to Educate and Activate (IDEA)
- 2 (Active Comparator): IE
  Interventions: Behavioral: Individual Education (IE)
- 3 (No Intervention): UC: Patients receive no research intervention.

INTERVENTIONS:
Behavioral: Interactive Dialogue to Educate and Activate (IDEA) — IDEA - patients receive group sessions totaling 8 hours, with an average of 10 patients per group, using conversation maps as a conduit to facilitate dialogue between providers and patients.
  Arms: 1
Behavioral: Individual Education (IE) — IE - patients receive 2 hours with a nurse educator and 1 hour with a dietitian.
  Arms: 2

SUMMARY:
Behavior change and self-efficacy are key for patients with diabetes to sustain blood sugar goals, but most care systems do not provide effective support to assist patients in successful ongoing self-management. After initial education, many programs are limited by allowable Medicare reimbursement for diabetes education which currently requires physician referral and cannot exceed two hours of training per year for a beneficiary, plus one hour of nutritional services. These services are usually provided either on an individual basis or occasionally through a traditional group class approach. For patients with established type 2 diabetes who are not achieving optimal glycemic control, we propose to develop and formally evaluate in a randomized trial a novel group experience to educate and motivate patients with established type 2 called IDEA, (Interactive Dialogue to Educate and Activate). This multi-site, randomized, prospective trial will randomize 621 patients with inadequately blood sugar control levels to one of 3 study groups: (1) IDEA - patients receive group sessions totaling 8 hours, with an average of 10 patients per group, using conversation maps as a conduit to facilitate dialogue between providers and patients (2) Individual Education (IE) - patients receive 2 hours with a nurse educator and 1 hour with a dietitian, and (3) Usual care (UC)- patients receive no research intervention. The primary analyses will involve mixed model regression to assess whether IDEA improves outcomes compared to IE and UC. Blood sugar level, blood pressure, and lipids will be evaluated 6 and12 months post-randomization and behavioral, emotional, and satisfaction outcomes through survey at baseline, 3, 6, 9 and 12 months. Depending on 12 month results, a longitudinal four year post intervention analysis is planned to assess sustainability of treatment effects and cost-effectiveness.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 Diabetes Mellitus

Exclusion Criteria:

* Gestational diabetes
* Type 1 Diabetes Mellitus

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 621 (Actual)
Dates: Start 2008-05-01 (Actual); Primary Completion 2010-03-01 (Actual); Study Completion 2011-07-01 (Actual)

PRIMARY OUTCOMES:
Program satisfaction, behavioral and emotional outcomes. | 3, 6, 9, 12 months after implementation of intervention

SECONDARY OUTCOMES:
Blood sugar level, blood pressure, lipids, cost, comorbidities. | 6, 12, 18, 24, 36, and 48 months after intervention

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
http://www.merck.com/clinical-trials/pdf/Merck%20Procedure%20on%20Clinical%20Trial%20Data%20Access%20Final_Updated%20July_9_2014.pdf
  http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Derived] Sperl-Hillen J, Beaton S, Fernandes O, Von Worley A, Vazquez-Benitez G, Parker E, Hanson A, Lavin-Tompkins J, Glasrud P, Davis H, Adams K, Parsons W, Spain CV. Comparative effectiveness of patient education methods for type 2 diabetes: a randomized controlled trial. Arch Intern Med. 2011 Dec 12;171(22):2001-10. doi: 10.1001/archinternmed.2011.507. Epub 2011 Oct 10. PMID 21986350